CLINICAL TRIAL: NCT05280106
Title: Comparison of Citrate Dialysate in Predilution and Postdilution Online Hemodiafiltration : Effect on Clot Formation and Adequacy of Dialysis in Hemodialysis Patients
Brief Title: Citrate Dialysate in Online Hemodialfiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080/64
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hemodiafiltration; Heparin; Haemodialysis; Citrate Reaction
Keywords: online hemodialfiltration; hemodialysis; citrate; adequacy of dialysis; heparin

STUDY DESIGN:
Intervention Model Description: One group interrupted times-series design (ITS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-dilution online hemodiafiltration (Experimental): The study was conducted for a 28-week period in two phases: For the first 12 weeks, all of the patients were subjected to CD with pre-dilution oL-HDF.After enrollment, all patients began a 2-week run-in period with conventional dialysis fluid containing acetate and the lowest dose of unfractionated heparin. The investigator titrated the heparin dose by reducing the dose step by step, 25% in each step, until the final minimal dose was achieved. The experimental study consisted of 3 phases, 4 weeks in each phase, and the phases were separated by 1-week washout periods. The second phase will run after finishing the first phase with the same protocol but with post-dilution online HDF.There will be 2 weeks washout period before starting this phase
  Interventions: Procedure: Pre-dilution online hemodiafiltration with citrate dialysate; Procedure: Post-dilution hemodiafiltration with citrate dialysate

INTERVENTIONS:
Procedure: Pre-dilution online hemodiafiltration with citrate dialysate — After enrollment, all patients began a 2-week run-in period with conventional dialysis fluid containing acetate and the lowest dose of unfractionated heparin. The investigator titrated the heparin dose by reducing the dose step by step, 25% in each step, until the final minimal dose was achieved. The experimental study consisted of 3 phases, 4 weeks in each phase, and the phases were separated by 1-week washout periods. Phase 1 used CD with 50% of the heparin dose of the baseline. Phases 2 and 3 used 25% heparin and no heparin, respectively. New dialyzers were introduced at the beginning of each phase and the heparin dose was resumed during the washout phase. The calcium concentration in the dialysis fluid was kept constant (1.5 mmol/L) to allow evaluation of the effect of CD on calcium balance
Procedure: Post-dilution hemodiafiltration with citrate dialysate — same protocol with post-dilution Ol-HDF in these same patients for the later 12 weeks.

SUMMARY:
Online hemodiafiltration (Ol-HDF) is increasingly being used for patients on chronic dialysis due to in its superiority compared with standard hemodialysis HDF. In addition to an excellent clearance of small molecules, oL-HDF has more advantages by providing both diffusion and convection modalities for an additional clearance of medium-size molecules. Furthermore, OL-HDF has been associated with not only better hemodynamic tolerance and biocompatibility , but may even include better survival.with reduction of proinflammatory cytokines and proinflammatory circulating cells , as well as with better control of B2MG levels .Ol-HDF is classified into 2 types according to the mode of addition of the substitution fluid: pre-dilution OL-HDF (pre-HDF) and post-dilution OL-HDF (post-HDF); Post-HDF was associated with significantly higher removal rates of β2-MG than HD. Postdilution HDF is the most effective way to maximize molecule clearance .Post-HDF was associated with significantly higher removal rate of α1-MG, and also significantly higher albumin leakage, than HD and pre-HDF. However, blood concentrations can be elevated using HDF, which can cause thrombosis. On the other hand, predilution HDF can resolve this problem but requires about three times more purified water than postdilution HDF and may not elicit maximal clearance.

DETAILED DESCRIPTION:
Heparin is the most routinely used anticoagulant in hemodialysis. However, it exposes the patient to the risk of bleeding complications and can induce thrombocytopenia. Furthermore, long-term use of heparin induces biological and clinical complications (osteoporosis, dyslipidemia, hyperkalemia) . Regional citrate anticoagulation is a good alternative to heparin use in hemodialysis for patients with increased bleeding risk , but its implementation in bicarbonate hemodialysis (BHD) is laborious and cumbersome: severe side effects can occur due to citrate metabolism and difficulties in adaptation of calcium infusion into the venous line .Therefore, the use of citrate as a dialysis buffer instead of acetate has proven a safe alternative to acetate-containing bicarbonate dialysis and on-line hemodiafiltration without significant hypocalcemia or clinically important coagulation issues.The aim of the present study is the comparison of the patency of the dialyzer ,the quality of life and blood parameters between pre and potdiltuiotn Ol-HDF with citrate dialysate (CD). No study to date has previously compared the use of citrate dialysate between these two modalities in oL-HDF.

ELIGIBILITY:
Inclusion Criteria:

* Stable condition
* Having been under HD for at least three months
* he vascular access should have blood flow ≥ 300 mL/min.

Exclusion Criteria:

* no heparin use during HD
* refusal to participate,
* intolerance or allergy to citrate
* concurrent infection
* poor life expectancy due to metastatic cancer, severe cirrhosis and AIDS.
* patients vascular access modification,
* patients affected by chronic liver disease, active neoplastic or inflammatory disease were excluded as well as patients receiving immunosuppressive or anti-inflammatory drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
clotting score between pre and post dilution online-hemodiafiltration | 28 weeks
  5 grades of clotting score, Grade 1;No or very little residual blood in the filters.Grade 1;Residual blood in less than 10% of the fibers. Grade 2; Residual blood 10-25%. Grade 3; Residual blood 25-50%.Grade 4 ,Residual blood > 50%

SECONDARY OUTCOMES:
quality of life between pre and post dilution online-hemodiafiltration | 28 weeks
  KDQOL-sf score;0-100.Higher scores reflect better quality of life
adequacy of dialysis between pre and post dilution online-hemodiafiltration | 28 weeks
  Kt/V
calcium level between pre and post dilution online-hemodiafiltration | 28 weeks
  serum calcium predialysis in midweek of each phase
phosphorus level between pre and post dilution online-hemodiafiltration | 28 weeks
  serum calcium predialysis in midweek of each phase
intact parathyroid level between pre and post dilution online-hemodiafiltration | 28 weeks
  serum parathyroid level in midweek of each phase

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Medicine ,Vajira hospital,Navamindradhiraj University, Bangkok
  - Faculty of Medicine ,Vajira Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Thaweethamcharoen T, Srimongkol W, Noparatayaporn P, Jariyayothin P, Sukthinthai N, Aiyasanon N, Kitisriworapan P, Jantarakana K, Vasuvattakul S. Validity and Reliability of KDQOL-36 in Thai Kidney Disease Patient. Value Health Reg Issues. 2013 May;2(1):98-102. doi: 10.1016/j.vhri.2013.02.011. Epub 2013 Mar 26. PMID 29702860
- [Result] Canaud B, Bosc JY, Leray H, Stec F, Argiles A, Leblanc M, Mion C. On-line haemodiafiltration: state of the art. Nephrol Dial Transplant. 1998;13 Suppl 5:3-11. doi: 10.1093/ndt/13.suppl_5.3. PMID 9623523
- [Result] Canaud B, Bragg-Gresham JL, Marshall MR, Desmeules S, Gillespie BW, Depner T, Klassen P, Port FK. Mortality risk for patients receiving hemodiafiltration versus hemodialysis: European results from the DOPPS. Kidney Int. 2006 Jun;69(11):2087-93. doi: 10.1038/sj.ki.5000447. PMID 16641921
- [Result] Guth HJ, Gruska S, Kraatz G. On-line production of ultrapure substitution fluid reduces TNF-alpha- and IL-6 release in patients on hemodiafiltration therapy. Int J Artif Organs. 2003 Mar;26(3):181-7. doi: 10.1177/039139880302600301. PMID 12703882
- [Result] Canaud B, Wizemann V, Pizzarelli F, Greenwood R, Schultze G, Weber C, Falkenhagen D. Cellular interleukin-1 receptor antagonist production in patients receiving on-line haemodiafiltration therapy. Nephrol Dial Transplant. 2001 Nov;16(11):2181-7. doi: 10.1093/ndt/16.11.2181. PMID 11682665
- [Result] Carracedo J, Merino A, Nogueras S, Carretero D, Berdud I, Ramirez R, Tetta C, Rodriguez M, Martin-Malo A, Aljama P. On-line hemodiafiltration reduces the proinflammatory CD14+CD16+ monocyte-derived dendritic cells: A prospective, crossover study. J Am Soc Nephrol. 2006 Aug;17(8):2315-21. doi: 10.1681/ASN.2006020105. Epub 2006 Jul 6. PMID 16825330
- [Result] Lin CL, Yang CW, Chiang CC, Chang CT, Huang CC. Long-term on-line hemodiafiltration reduces predialysis beta-2-microglobulin levels in chronic hemodialysis patients. Blood Purif. 2001;19(3):301-7. doi: 10.1159/000046958. PMID 11244190
- [Result] Kurihara Y, Hosoya H, Kishihara R, Yoshinaga M, Iwadate Y, Yamauchi F, Saito T, Sakurai K. Comparison of the effects of pre-dilution and post-dilution online hemodiafiltration on the levels of inflammatory markers, lymphocytes, and platelets. J Artif Organs. 2022 Mar;25(1):59-65. doi: 10.1007/s10047-021-01281-5. Epub 2021 Jun 14. PMID 34128110
- [Result] Tsuchida K, Minakuchi J. Clinical benefits of predilution on-line hemodiafiltration. Blood Purif. 2013;35 Suppl 1:18-22. doi: 10.1159/000346221. Epub 2013 Feb 25. PMID 23466373
- [Result] Hottelart C, Achard JM, Moriniere P, Zoghbi F, Dieval J, Fournier A. Heparin-induced hyperkalemia in chronic hemodialysis patients: comparison of low molecular weight and unfractionated heparin. Artif Organs. 1998 Jul;22(7):614-7. doi: 10.1046/j.1525-1594.1998.06204.x. PMID 9684701
- [Result] Aniort J, Petitclerc T, Creput C. Safe use of citric acid-based dialysate and heparin removal in postdilution online hemodiafiltration. Blood Purif. 2012;34(3-4):336-43. doi: 10.1159/000345342. Epub 2013 Jan 9. PMID 23306782